CLINICAL TRIAL: NCT04988997
Title: A Phase 2, Double-Blind, Double-Dummy, Placebo-Controlled, Multicenter Study of the Efficacy, Safety, and Tolerability of Vurolenatide in Adult Patients With Short Bowel Syndrome
Brief Title: VIBRANT Study of Vurolenatide in Adult Patients With Short Bowel Syndrome.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial terminated by Sponsor
Sponsor: 9 Meters Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMSBS01-002
Record Dates: First submitted 2021-07-19; First posted 2021-08-04 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Double-Blind, Double-Dummy, Placebo-Controlled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind, Double-Dummy, Placebo-Controlled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Vurolenatide 50 mg/PBO (Active Comparator): 50 mg biweekly SC administration, PBO alternate weeks
  Interventions: Drug: Vurolenatide 50mg/PBO
- Vurolenatide 100 mg/PBO (Active Comparator): 100 mg biweekly SC administration, PBO alternate weeks
  Interventions: Drug: Vurolenatide 100mg/PBO
- Vurolenatide 50/50 mg (Active Comparator): 50 mg weekly SC administration
  Interventions: Drug: Vurolenatide 50/50 mg
- Placebo (Placebo Comparator): PBO - weekly SC administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vurolenatide 50mg/PBO — Vurolenatide - 50 mg biweekly SC administration, PBO alternate weeks
  Arms: Vurolenatide 50 mg/PBO
Drug: Vurolenatide 100mg/PBO — Vurolenatide - 100 mg biweekly SC administration, PBO alternate weeks
  Arms: Vurolenatide 100 mg/PBO
Drug: Vurolenatide 50/50 mg — Vurolenatide - 50 mg weekly SC administration
  Arms: Vurolenatide 50/50 mg
Drug: Placebo — PBO - weekly SC administration
  Arms: Placebo

SUMMARY:
A Study of Vurolenatide in Adult Patients with Short Bowel Syndrome.

DETAILED DESCRIPTION:
A Phase 2 study of Vurolenatide in adult patients with SBS. Patients were planned to be dosed in four treatment groups with placebo and/or active Vurolenatide. The study is 13 weeks (3 weeks screening, 4 weeks SC study drug administration, and 6 weeks of follow up). Safety and efficacy will be analyzed.

ELIGIBILITY:
Key Inclusion Criteria:

Criteria for patient inclusion in this study are as follows:

1. Male and female adults with SBS secondary to surgical resection of small intestine
2. 18-75 years of age at the time of screening.
3. Female patients must be postmenopausal (at least 2 years prior to dosing) or surgically sterile or agree to use an acceptable form of birth control from screening until 30 days after last dose. If oral contraceptives are used, patients must have been on a stable dose for ≥6 months.
4. Male patients must agree to use an acceptable form of birth control during the study and for 30 days after the last dose. Male patients should not donate sperm for 90 days after last dose.
5. At least 6 months since last surgical bowel resection.
6. Patients may be on Parenteral Support [PS] (nutrition and/or fluid and electrolytes for at least some of their nutritional needs).
7. If on PS, stable administration of PS volume for 1 month (±20% vol) prior to enrollment [stable administration of PS volume confirmed by Medical Monitor].
8. Able to ingest solid or semi-solid foods and drink.

Key Exclusion Criteria:

Criteria for exclusion from participation in this study are presented below.

1. Pregnancy or lactation
2. Body mass index at screening <18 or >30 kg/m2
3. Clinically significant intestinal adhesions and/or chronic abdominal pain that can interfere with the conduct of the study
4. Active Crohn's disease or IBD (as evaluated by standard procedures employed by the investigator/institution). If in remission, must be ≥12 weeks of remission prior to screening
5. Inflammatory bowel disease patients who have NOT been on a stable drug treatment regimen for at least the past 3 months prior to screening
6. Visible blood in the stool within the last 3 months
7. Known heart failure or active coronary disease
8. Alcohol or drug abuse within the last 12 months by history, or a disqualifying positive urine drug test at screening.
9. Inadequate renal function as defined by serum creatinine <0.7 or >1.3 mg/dL (in men) and <0.6 or >1.1 mg/dL in women.
10. Personal or family history of medullary thyroid cancer.
11. History of pancreatitis
12. Any use of growth hormone, or growth factors such as native GLP-2 or GLP-2 analog (teduglutide) within the last 3 months
13. Use of antibiotics within the last 30 days
14. Patient not capable of understanding or not willing to adhere to the study visit schedules and other protocol requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
24hr total stool output volume | 10 weeks (including 6 weeks follow up)
  The primary outcome measure is 24hr total stool output volume over the double-blind treatment period compared to baseline.

SECONDARY OUTCOMES:
Assess the safety and tolerability of vurolenatide | 10 weeks (including 6 weeks follow up)
  Assessment of Adverse events - The frequency of spontaneously reported AEs will be assessed for each treatment group separately by System Organ Class and Preferred Term; and vital signs, physical examination results, clinical laboratory tests results will be evaluated.
To assess change from Baseline in Quality of Life | 10 weeks (including 6 weeks follow up)
  Change from baseline in Quality of Life as measured by the SF-36 instrument over the double-blind treatment period
To assess the change from baseline in Patient Global Impression | 10 weeks (including 6 weeks follow up)
  Change from baseline in patient reported global SBS improvement over the double-blind treatment period

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Research Site, Gainesville, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Boston, Massachusetts
  - Research Site, Omaha, Nebraska
  - Research Site, Durham, North Carolina
  - Research Site, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No